CLINICAL TRIAL: NCT02296060
Title: Evaluation of Exercise Tolerance During Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 6MWT pregnancy
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6 minutes walking test (Experimental)
  Interventions: Procedure: 6 minutes walking test

INTERVENTIONS:
Procedure: 6 minutes walking test

SUMMARY:
To evaluate the exercise tolerance during pregnancy and after thanks the 6MWT

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* healthy women

Exclusion Criteria:

* BMI (before pregnancy) > 25
* complication with their pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
6 minutes walking test | after 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Woluwé-Saint-Lambert, Belgium